CLINICAL TRIAL: NCT04954573
Title: Pilot Study on the Treatment With Water-filtered Infrared-A (wIRA) Radiation in Patients With Morphea and Sclerotic Graft-versus-host Disease
Brief Title: Study on the Treatment With Water-filtered Infrared-A (wIRA) Radiation in Patients With Morphea and Sclerotic Graft-versus-host Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was prematurely terminated due to recruitment difficulties.
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30-387 ex 17/18
Record Dates: First submitted 2021-06-09; First posted 2021-07-08 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Morphea (Circumscribed Scleroderma); Sclerotic Graft-versus-host Disease (GVHD)
MeSH Terms: conditions — Scleroderma, Localized

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morphea (Other)
  Interventions: Radiation: infrared-A (wIRA)
- Sclerotic graft-versus-host disease (GVHD) (Other)
  Interventions: Radiation: infrared-A (wIRA)

INTERVENTIONS:
Radiation: infrared-A (wIRA) — Local-water filtered infrared-A (wIRA) irradiation

SUMMARY:
This is a prospective, intra-individual comparative study to evaluate the effectiveness of local-water filtered infrared-A (wIRA) irradiation (applied by Hydrosun® radiator 750 for radiation at the clinic, or Hydrosun® 575home for home treatment) in patients with morphea or sclerotic GVHD (Graft-versus-host Disease). The purpose of the study is to determine whether wIRA irradiation can reduce fibrotic skin alterations in circumscribed scleroderma (morphea) or chronic graft versus host disease. wIRA irradiation is applied for 30 minutes 3 times per week for 20 weeks to a diseased skin area and a lesional skin on contralateral body site remains untreated. A total of 22 patients (20 evaluable patients with an expected drop-out rate of 10%) are to be included in this study. Group A: 11 patients with plaque morphea Group B: 11 patients with sclerotic GVHD.

DETAILED DESCRIPTION:
A sclerotic plaque or area of skin on the right side of the body and contralaterally on the left half of the body (each maximum size: 25 cm in diameter, corresponding to the radiation field of the Hydrosun® heater 750) is selected. The assignment of one side of the body to irradiation or non-irradiation is randomized (using the MedUni Graz randomizer). The plaque randomized for irradiation is irradiated on 3 days a week for 30 minutes each time. The treatment period extends over 20 weeks, the total number of radiation treatments is therefore 60. If the patients cannot come to the radiation treatment, home therapy can be carried out according to the same treatment scheme. The radiation at the clinic is carried out with a Hydrosun® lamp 750, the home treatment with the Hydrosun® 575home (Hydrosun Medizintechnik GmbH, Mauchener Str. 14, D-79379 Muellheim, Germany). The radiation intensity at the distance of 33 cm between the device and the skin surface standardized by a distance rod is 200 mW / cm2 (visible light 50 mW / cm2, infrared A 150 mW / m2). The contralateral plaque or skin area of comparable clinical characteristics and duration of existence was included as an unirradiated control. Target and control areas will be photo-documented in the course of the study. Before the first irradiation, after the 30th and after the 60th irradiation, the skin thickness and hardness of the target and control regions are measured by a blinded examiner and the skin status including mRSS (Rodnan skin score) is recorded. In addition, at the beginning and at the end of the study, the patient's assessment of the effect (PGIC scale) and tolerability of the therapy is asked. Any side effects of the irradiation are continuously documented.

ELIGIBILITY:
Inclusion Criteria:

* Morphea
* Sclerotic graft-versus-host disease (GVHD)

Exclusion Criteria:

* Inability to cope with the treatment plan
* Pregnant or breastfeeding women and women of childbearing potential without effective contraception

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-02-13 (Actual); Study Completion 2024-02-13 (Actual)

PRIMARY OUTCOMES:
Intensity of skin sclerosis | 20 weeks
  as determined by a high-frequency ultrasound device with a 22 MHz applicator

SECONDARY OUTCOMES:
Assessment of skin Score | 20 weeks
  determined by modified Rodnan Skin Score (mRSS) (range, 0 to 51 )
Assessment of skin hardness | 20 weeks
  as determined by durometer
Assessment of range of motions | 20 weeks
  as measured by the range of motions in the presence of contractures (range, 0 to 90 degree)
Grade of patient satisfaction | 20 weeks
  as determined by Patients' Global Impression of Change (PGIC) scale (range, 0 to 7)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wolf, MD, Principal Investigator — Medical University of Graz
Locations (2):
- Austria (2):
  - Department of Dermatology, Medical University of Graz, Graz, Styria
  - Department of Dermatology, Medical University of Vienna, Vienna

IPD SHARING:
Plan to Share IPD: Undecided